CLINICAL TRIAL: NCT03194555
Title: Randomized, Double-Blind, Study to Assess Low-Dose Naltrexone and Acetaminophen Combination in the Prevention of Episodic Migraine in Adults
Brief Title: The Preventive Treatment of Migraine With Low-Dose Naltrexone and Acetaminophen Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allodynic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANODYNE-3
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Migraine With or Without Aura
Keywords: Innate Immune System; Cytokines; Cox-2; Headache; Migraine; Migraine Prevention
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Dose Naltrexone and Acetaminophen Combination (Experimental)
  Interventions: Drug: Low-Dose Naltrexone and Acetaminophen Combination
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-Dose Naltrexone and Acetaminophen Combination — Twice daily
  Arms: Low-Dose Naltrexone and Acetaminophen Combination
Drug: Placebo — Twice daily
  Arms: Placebo

SUMMARY:
The Preventive Treatment of Migraine with Low-Dose Naltrexone and Acetaminophen Combination: A Small, Randomized, Double-Blind, and Placebo-Controlled Clinical Trial with an Open-Label Extension for None-Responders

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a male or a female 18 years of age or older.
2. History of migraine with or without aura according to the International Classification of Headache Disorders (ICHD)-3rd edition (beta version) for at least one-year with onset of migraine prior to 50 years of age.
3. Migraine-associated nausea with ≥half of migraine attacks.
4. 5-8 migraine/probable migraine headache days on average per month in the three months prior to Visit 1 and during the Baseline Period.
5. The patient agrees to refrain from taking opiate medications from Visit 1 to 7 days after the last dose of the study drug.
6. The patient is able to complete study questionnaires, comply with the study requirements and restrictions, and willing to provide written informed consent and authorize HIPAA.
7. The patient has been taking a stable dose of a medication with migraine prevention potential for at least 3 month prior to the screening visit and agrees to not start, stop, or change dosage of any medication with migraine prevention potential during the study period. (E.g., beta-blockers, calcium channel blockers, tricyclic antidepressants, anticonvulsants, selective serotonin re-uptake inhibitors (SSRIs), serotonin-norepinephrine re-uptake inhibitors (SNRIs), magnesium or riboflavin supplements at high doses, herbal preparations (e.g. feverfew or St. john's wort)), Botulinum toxin must be discontinued one year prior to Visit 1.
8. The patient agrees to forgo any elective surgery for the duration of the study.
9. The female patient who is premenopausal or postmenopausal less than 1 year, or have not had surgical sterilization (i.e., tubal ligation, partial or complete hysterectomy) must have a negative urine pregnancy test, be non-lactating, and commit to using 2 methods of adequate and reliable contraception throughout the study and for 28 days after taking the last dose of the study drug (e.g., barrier with additional spermicidal, intra-uterine device, hormonal contraception). Male patients must be surgically sterile or commit to the use of 2 different methods of birth control during the study and for 28 days after the study.

Exclusion Criteria:

1. Usage of acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDs) ≥15 days/month, or ergotamine and triptans >10 days/month, or opioids and barbiturates >2 days/month in the 3 months prior to Visit 1 or during the Baseline Period.
2. Tension-type-like, and/or migraine-like headache on ≥15 days per month in the 3 months prior to Visit 1 or during the Baseline Period. Diagnosis of chronic migraine, cluster headache or neurologically complicated migraine (hemiplegic, basilar, retinal, ophthalmoplegic migraine).
3. Regular use of the following medications for any reason: acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), antipsychotic drugs, monoamine oxidase inhibitors, benzodiazepines, sleep medications, muscle relaxants, anti-emetic medications, blood thinning medications (e.g., warfarin or heparin), cannabinoids, or botulinum toxin to head and neck regions. Low-dose aspirin for cardiovascular disease prophylaxis is permitted.
4. Confounding painful conditions, (e.g. fibromyalgia, chronic low back pain, complex regional pain syndrome, etc.).
5. Diagnosis of any concurrent medical or psychiatric condition; this includes, chronic unstable debilitating diseases such as Parkinson's disease, multiple sclerosis, cancer, significant renal impairment, significant hepatic impairment, etc.
6. The patient has a history or diagnosis of moderate-to-severe hepatic or renal impairment (>2 × the upper limit of normal [ULN] for alanine transaminase or aspartate transaminase. ≥1.5 × ULN for alkaline Phosphatase, bilirubin, BUN, or creatinine). (Patients with elevated bilirubin level due to Gilbert's syndrome are allowed).
7. The patient has a history within the previous 5 years of abuse of any drug, prescription, illicit, or alcohol.
8. The Female patient is pregnant, actively trying to become pregnant, or breast-feeding. The Male patient is not practicing 2 different methods of birth control with their partner during the study, and for 28 days after the investigational drug last dose or will not remain abstinent during the study, and for 28 days after the last dose.
9. The patient has known-allergy to any of the components of the investigational drug.
10. Participation in another study with an investigational drug within 30 days before Visit 1 or during the study.
11. Use of emergency care treatment more than 3 times in the previous 6 months.
12. The patient is in the opinion of the investigator, is unsuitable to participate in this study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Toledano, M.D., Principal Investigator — Allodynic Therapeutics, Inc
Locations (1):
- Annette Toledano, M.D., North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment was conducted in a single site in Miami, Florida.
Period: Overall Study
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all treated participants (all enrolled participants who took the study drug).
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (14.3) | 39 (10.4) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 5 | 11
  African American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Monthly Migraine Days (MMD) From Baseline to the Last 28 Days of Treatment Period.
Description: Migraine with or without aura is defined according to the International Classification of Headache Disorders (ICHD)-3rd edition (beta version). Migraine headaches must be moderate or severe and lasting ≥30 minutes. When the patient falls asleep during migraine and wakes up without it, duration of the attack is reckoned until the time of awakening).
Time Frame: From the 28-day baseline period to the last 28 days of the 84-days double-blinded treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
days | -5.67 (3.2) | -3.5 (5.56)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.4267, Chi-squared; Risk Difference (RD) = -2.17, 95% CI 2-sided [-3.67 to 8.01]

2. Secondary Outcome: The Number of Participants With More Than 50% Improvement in the Mean Monthly Migraine Days (MMDs)
Description: MMD stands for change in Monthly Migraine Days from 28-day baseline to the last 28 days of the double-blind treatment period
Time Frame: From the 28-day baseline period to the last 28 days of the 84-days double-blinded treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 4 | 2
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.268, Chi-squared; Risk Difference (RD) = 2, 95% CI 2-sided [-18.46 to 66.83]

3. Secondary Outcome: The Number of Participants With More Than 75% Improvement in the Mean Monthly Migraine Days (MMDs)
Time Frame: From the28-day baseline period to the last 28 days of the 84-day treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 4 | 1
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.0926, Chi-squared; Risk Difference (RD) = 3, 95% CI 2-sided [-17.2 to 67.4]

4. Secondary Outcome: The Number of Participants With 100% Improvement in Mean MMD in the Last 28 Days Double-blinded Treatment Period.
Time Frame: From the 28-day baseline period to the last 28 days of the 84-day treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 3 | 1
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.2894, Chi-squared; Risk Difference (RD) = 2, 95% CI 2-sided [-17.2 to 67.4]

5. Secondary Outcome: Mean Monthly Acute Migraine Medication Treatment Days Change From Baseline to Last 28 Days of Treatment
Time Frame: From the 28-day baseline period to the last 28 days of the 84-day treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
days
  Baseline acute number of migraine medication treatment days | 7.67 (2.07) | 8.67 (3.5)
  Acute migraine medication treatment days in last 28 days of treatment period | 2.67 (4.32) | 5.5 (3.27)
  change in monthly acute migraine medication treatment days baseline to last 28 days of treatment | -5 (5.37) | -3.17 (5.49)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.5724, Chi-squared; Risk Difference (RD) = -1.83, 95% CI 2-sided [-5.1557 to 8.8157]

6. Secondary Outcome: The Change in HIT-6 From Baseline to Last 28 Days of Treatment
Description: HIT-6 - headache impact test - was designed to provide a global measure of adverse headache impact. Score range is 36-78, Score ≥ 60 - a very severe impact on life, scored ≤ 49 little to no impact on life. The percent responders were calculated as follows: the change from baseline score divided by the score at the baseline minus 36.
Time Frame: From the 28-day baseline period to the last 28 days of the 84-day treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
score
  Baseline (Randomization visit) mean HIT-6, score | 68.5 (5.68) | 68.83 (5.27)
  HIT-6 in last 28 days of treatment, score | 47.83 (17.69) | 58 (12.08)
  The change in HIT-6 from baseline to last 28 days of treatment, score | -20.67 (19.08) | -10.83 (12.98)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.2998, Chi-squared; Risk Difference (RD) = -9.84, 95% CI 2-sided [-11.15 to 30.83]

7. Other Pre Specified Outcome: The Change in Mean PIRS-20 From Baseline to Last 7 Days of Treatment.
Description: Average of PIRS-20, (0-60 = higher with difficulty with sleep)
Time Frame: From baseline to month 3 of the treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug,
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
score
  Baseline (Randomization visit) mean PIRS-20, score | 32.67 (16.97) | 31.83 (7.03)
  PIRS-20 in last week of treatment period, score | 10 (19.32) | 20.83 (14.39)
  The change in PIRS-20 from baseline to last week of treatment, score | -22.67 (22.64) | -11 (8.92)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.2673, Chi-squared; Risk Difference (RD) = -11.67

8. Other Pre Specified Outcome: The Number of Participants Who Had an Improvement in Patient Global Impression of Change (PGIC) at End of Treatment
Time Frame: From baseline to month 3 of the treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  PGIC, Change≥2 points, (%) | 4 | 2
  PGIC, Change=3 points, (%) | 4 | 2

9. Other Pre Specified Outcome: The Number of Participants Reporting Patients' Satisfaction Level
Time Frame: From baseline to month 3 of the treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  Satisfied or very satisfied (level 2 or 3) | 4 | 2
  Very satisfied (level 3) | 4 | 2

10. Other Pre Specified Outcome: Mean Monthly Migraine Hours Change From Baseline to Last 28 Days of Treatment
Time Frame: From baseline to month 3 of the treatment period.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Hours
  Baseline, hours | 70.78 (47.6) | 54.44 (36.21)
  Monthly migraine hours in last 28 days of treatment, hours | 24.65 (35.23) | 37.07 (38.05)
  The change in monthly migraine hours from baseline to last 28 days of treatment, hours | -46.13 (59.44) | -17.37 (41.11)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.3527, Chi-squared; Risk Difference (RD) = 28.76, 95% CI 2-sided [-94.5005 to 36.9805]

11. Other Pre Specified Outcome: Change in at Least Moderate Migraine Days in Treatment
Time Frame: From baseline to month 3 of the treatment period
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
days
  Mean monthly at least moderate Headaches days at baseline | 8.33 (2.73) | 9 (2.45)
  Mean at least moderate migraine days in the last 28 days of the treatment period | 3.67 (5.57) | 6.17 (4.54)
  The change in at least moderate migraine days from baseline to the last 28 days of treatment period | -4.78 (4.42) | -2.83 (5.74)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.5246, Chi-squared; Risk Difference (RD) = -1.95

12. Other Pre Specified Outcome: The Number of Participants Who Achieved the Percentage of Response in at Least Moderate Migraine Days Baseline to Last 28 Days of Treatment
Time Frame: From baseline to month 3 of the treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  ≥50% | 4 | 2
  ≥75% | 4 | 1
  ≥90% | 3 | 1
  100% | 3 | 1

13. Other Pre Specified Outcome: Mean Severe Headache Days Change From Baseline to Last 28 Days of Treatment
Time Frame: From baseline to month 3 of the treatment period.
Population: Modified intent to treat (mITT) participants included all randomized participants who took study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
Number analyzed (Participants) | 6 | 6
days
  Mean monthly severe headaches days at baseline | 4.83 (1.72) | 4.33 (2.88)
  Mean severe headache days in the last 28 days of the treatment period | 2.67 (3.93) | 2.5 (3.02)
  The change in severe headache days from baseline to the last 28 days of the treatment period | -2.17 (2.79) | -1.83 (3.87)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone and Acetaminophen Combination vs Placebo; Test type: Superiority; p = 0.8649, Chi-squared; Risk Difference (RD) = 0.34

ADVERSE EVENTS:
Time Frame: One month follow-up after 3 months of treatment
Description: The safety population included all the 12 randomized patients who took the study drug (ITT).
Arm/Group | Low-Dose Naltrexone and Acetaminophen Combination | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-Dose Naltrexone and Acetaminophen Combination (N=6) | Placebo (N=6)
Dry Mouth (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 | 0
Heavy Breathing (General disorders) | 1 | 1
Nausea (General disorders) | 1 | 0
Palpitations (General disorders) | 1 | 0
Somnolence (General disorders) | 1 | 1
Vomiting (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03194555/Prot_SAP_000.pdf